CLINICAL TRIAL: NCT03779269
Title: Effect of Preksha Meditation (Green Color and Buzzing Meditation) on Cognitive Abilities and Pulmonary Function in Students With a Control Group
Brief Title: Effect of Preksha Meditation on Cognitive Abilities and Pulmonary Function in Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Orlando Regional Medical Center (Other)
Collaborators: Florida International University (Other)
Responsible Party: Principal Investigator, Devendra Mehta, Director Translational Research laboratory, Orlando Regional Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-13-0045-CR03
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Inattention and Memory; Affect
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Intervention Model Description: prospective convenience controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- color meditation (Experimental): only color meditation
  Interventions: Other: meditation
- Sound meditation (Experimental): Only sound mediation
  Interventions: Other: meditation
- Color and sound combined meditation (Experimental): Combined group
  Interventions: Other: meditation
- Control group (No Intervention): Only control group

INTERVENTIONS:
Other: meditation — meditation effect assessment using assessment tools.
  Arms: Color and sound combined meditation; Sound meditation; color meditation

SUMMARY:
The goal of this project is to assess impact of an 8 week course of Preksha Meditation (combination of Green color and buzzing sound meditation), in a group of college students to assess potential benefits to their pulmonary function, cognitive ability (immediate recall, attention), and happiness.

DETAILED DESCRIPTION:
Preksha Meditation Research: The goal of this project is to assess impact of an 8 week course of Preksha Meditation (combination of Green color and buzzing sound meditation), in a group of college students to assess potential benefits to their pulmonary function, cognitive ability (immediate recall, attention), and happiness. The investigators will compare the data received from prior study to analyze their performance before and after. The investigators will also compare this data with control group data, to assess potential improvements as a benchmark. Analyse the EEG data to investigate its impact on brain. Further analyze their blood cells if they show any epigenetic changes. Data analysis team will be blinded for no identifiers are available.

METHOD AND PROCEDURES:

The data analysis will be undertaken by experts and will be blinded. The data currently is only de-identified.

The data which is already collected from the research "Effect of Preksha Meditation (Green color and Buzzing Meditation) on Cognitive Abilities and Pulmonary Function in Students with a Control Group" will be analyzed. The data is related to students having practiced minimum 3 guided 25 minute sessions per week in a controlled environment. The control group did not meditate for those weeks when they enrolled in the program.

The intervention the subjects received was as follows:

Experimental group 3 days per week Sessions: 5 minutes: Relaxation and Review of Meditation Practices 10 minutes: Mahapraan Meditation 10 minutes: Green color meditation Begin in stages

* 0 - 2 Weeks: Teach technique and carry out 15 minutes meditation sessions.
* 2 - 9 Weeks: Increment meditation sessions to a length of 25 minutes. 5 minutes: Review of meditation experience and collection of information

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* No prior experience in meditation

Exclusion Criteria:

* Prior experience with meditation.

  * health issues.
  * Alcohol
  * Smoking.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2017-05-14 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
Cognitive skills assessment using Connor's CPT test | 8 weeks
  Affect, short term memory, inattention,

SECONDARY OUTCOMES:
Pulmonary function using actual lung capacity test | 8 weeks
  Spirometry
Transcriptomics and epigenetics | 8 weeks
  Upregulation and transcriptional profiling using fold change

CONTACTS AND LOCATIONS:
Overall Officials: Devendra Mehta, M.D., M. SC., Principal Investigator — Head, Translational Research
Locations (2):
- United States (2):
  - Florida International University, Miami Beach, Florida
  - Orlando Regional Medical Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
De-identified summary data

REFERENCES:
- [Background] Mehta S, Mehta V, Mehta S, Shah D, Motiwala A, Vardhan J, Mehta N, Mehta D. Multimodal behavior program for ADHD incorporating yoga and implemented by high school volunteers: a pilot study. ISRN Pediatr. 2011;2011:780745. doi: 10.5402/2011/780745. Epub 2011 Aug 11. PMID 22389788
- [Background] Pragya SU, Cordoba G, Chiu R, Mehta N, Johnson P, Mehta DI, Mehta N. Can The Cognitive Parameters Of College Students With Learning Disabilities Benefit From Using Mahapraan, A Breathing Based Preksha Meditation. Journal of College Teaching & Learning 2014; 11, 4 Epub
- [Derived] Pragya SU, Pragya SC, Griswold AJ, Gu E, Mehta ND, Uddin P, Veeramachaneni P, Mehta N, Mehta D, Abomoelak B. Preksha Dhyana Meditation Effect on the DNA Methylation Signature in College Students. J Integr Complement Med. 2023 Apr;29(4):224-233. doi: 10.1089/jicm.2022.0713. Epub 2023 Feb 7. PMID 36749149
- [Derived] Pragya SU, Mehta ND, Abomoelak B, Uddin P, Veeramachaneni P, Mehta N, Moore S, Jean-Francois M, Garcia S, Pragya SC, Mehta DI. Effects of Combining Meditation Techniques on Short-Term Memory, Attention, and Affect in Healthy College Students. Front Psychol. 2021 Mar 5;12:607573. doi: 10.3389/fpsyg.2021.607573. eCollection 2021. PMID 33746830